CLINICAL TRIAL: NCT03284593
Title: Prognostic Factors and the Impact of Various Management of Acute Myeloid Leukemia in Real Life Condition at Toulouse and Bordeaux University Hospital
Brief Title: Prognostic Factors and the Impact of Various Management of Acute Myeloid Leukemia in Real Life Condition
Acronym: LAM-BDD
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 14 7344 03
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intensive chemotherapy group: patients treated with intensive chemotherapy
  Interventions: Drug: intensive chemotherapy
- Azacitidine group: patients treated with azacitidine
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: intensive chemotherapy
  Groups: intensive chemotherapy group
Drug: Azacitidine
  Groups: Azacitidine group

SUMMARY:
The treatment of older patients with acute myeloid leukemia that is secondary to previous myelodysplastic syndrome, myeloproliferative neoplasm, or prior cytotoxic exposure remains unsatisfactory. We compared patients treated with intensive chemotherapy or azacitidine within two centres.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute myeloid leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of acute myeloid leukemia between 2000 and 2014 in 2 hospitals in South of France
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2014-12; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  Survival times

CONTACTS AND LOCATIONS:
Overall Officials: Christian RECHER, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital Bordeaux, Bordeaux
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No